CLINICAL TRIAL: NCT06326840
Title: Predictive Models of Clinical Efficacy and Adverse Reactions of Antipsychotic Treatment
Brief Title: Clinical Efficacy and Adverse Reactions of Antipsychotic Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University Hospital (Other)
Collaborators: Taipei Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 98107
Record Dates: First submitted 2024-02-23; First posted 2024-03-22 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2010-05

CONDITIONS: Metabolic Disturbance; Hyperprolactinemia; Schizophrenia
Keywords: schizophrenia; olanzapine; metabolic disturbance; prolactin
MeSH Terms: conditions — Hyperprolactinemia; Schizophrenia | interventions — Metformin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- metformin intervention (Experimental): All participants were administered 1500 mg/day of metformin for eight weeks.
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Metformin — All participants were administered 1500 mg/day of metformin for eight weeks. The trial design is single-group with no masking.

SUMMARY:
The goal of this clinical trial is to explore the potential of metformin in managing olanzapine-induced metabolic disturbance and hyperprolactinemia in patients with schizophrenia. The main questions it aims to answer are:

1. The effect of metformin on olanzapine-induced metabolic disturbance
2. The effect of metformin on olanzapine-induced hyperprolactinemia

Participants will receive metformin 1500 mg/day for 8 weeks and assessments every 2 weeks.

DETAILED DESCRIPTION:
The study was conducted in an inpatient setting, with the dosage of olanzapine remaining consistent throughout the study duration. All participants were administered 1500 mg/day of metformin for eight weeks. Vital signs were measured daily. Physical and neurological examinations were carried out on a weekly basis. Every two weeks, all participants underwent an assessment for general psychopathology. Blood samples were collected in the morning after an overnight fast at the beginning of the study and then every two weeks following the commencement of metformin treatment. Serum prolactin levels were determined through electrochemiluminescence immunoassays. Fasting serum levels of glucose, total cholesterol, high-density lipoprotein cholesterol (HDL-C), low-density lipoprotein cholesterol (LDL-C), and triglycerides were measured using enzymatic colorimetric assays. Serum insulin and leptin levels were measured using electrochemiluminescence immunoassay kits.

ELIGIBILITY:
Inclusion Criteria:

* aged between 18 and 60 years
* diagnosed with schizophrenia under the Diagnostic and Statistical Manual of Mental Disorders-fourth edition criteria
* had been consistently treated with a stable dose of olanzapine for a minimum of three months

Exclusion Criteria:

* Exclusion criteria encompassed any mental disorder other than schizophrenia, ongoing substance abuse, and medical conditions that could interfere with glucoregulatory and endocrine assessment such as diabetes mellitus and other endocrine disorders. Additionally, severe cardiovascular, hepatic, or renal diseases, malignancy, epilepsy, and pregnancy were also reasons for exclusion.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2010-05-31 (Actual); Primary Completion 2011-06-10 (Actual); Study Completion 2011-06-10 (Actual)

PRIMARY OUTCOMES:
Glucose level | 8 weeks
  Glucose level was measured every 2 weeks.
prolactin level | 8 weeks
  Prolactin level was assessed every 2 weeks.
Insulin level | 8 weeks
  insulin level was measured every 2 weeks
low-density lipoprotein cholesterol (LDL-C) level | 8 weeks
  LDL-C level was measured every 2 weeks
high-density lipoprotein cholesterol (HDL-C) level | 8 weeks
  HDL-C level was measured every 2 weeks
cholesterol level | 8 weeks
  cholesterol level was measured every 2 weeks
triglycerides level | 8 weeks
  triglycerides level was measured every 2 weeks
leptin level | 8 weeks
  leptin level was measured every 2 weeks

SECONDARY OUTCOMES:
Clinical Global Impression scale | 8 weeks
  The clinical global impression scale was applied every 2 weeks. The clinical global impression scale is a 7-point scale that requires the clinician to rate the severity of the patient's illness at the time of assessment. The clinical global impression scale is rated from 0 (normal, not at all ill) to 7 (Among the most extremely ill patients).

CONTACTS AND LOCATIONS:
Overall Officials: Mong-Liang Lu, MD, Principal Investigator — Taipei Meidcal University-Wan Hospital
Locations (1):
- Taipei Medical University-Wan Fang Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No